CLINICAL TRIAL: NCT01229631
Title: The Effect of Daily Dietary Intake of Dried Juice Concentrates of Fruit, Vegetables and Berries (Juice Plus+) Upon Periodontal Outcomes in Chronic Periodontitis: A Multicentre Randomised Controlled Trial
Brief Title: The Effect of Daily Dietary Intake of Dried Juice Concentrates of Fruit, Vegetables and Berries Upon Outcomes of Chronic Periodontitis
Acronym: ENURGISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Community Healthcare NHS (Other Government)
Collaborators: University of Wuerzburg (Other); Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Professor I Chapple, Professor (PI to study), Birmingham Community Healthcare NHS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MULTI-NSA-10-001
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; Dietary supplementation
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: longitudinal, randomised, block stratified (for smoking), double-blind, 2-arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation with non-active (Placebo Comparator): Subjects will be supplemented with placebo capsules (3 capsules am & 3 capsules pm)
  Interventions: Dietary Supplement: Placebo non active capsules
- Dietary supplementation with Juice plus+ (Active Comparator): Subjects will be supplemented with Juice plus+ capsules (3 capsules am & 3 capsules pm)
  Interventions: Dietary Supplement: Juice plus+

INTERVENTIONS:
Dietary Supplement: Juice plus+ — Subjects in active group will be supplemented with Juice plus+ capsules (3 in the morning and 3 in the evening, for 3 months)
  Arms: Dietary supplementation with Juice plus+
Dietary Supplement: Placebo non active capsules — Subjects will take non-active placebo capsules (3 in the morning and 3 in the evening, for 3 months)
  Arms: Supplementation with non-active

SUMMARY:
The objective of this study is to determine whether enhanced micronutrient intake in the form of fruit, vegetable and berry juice powder (FVB) concentrate, improves clinical outcomes in chronic periodontitis patients prior to standard non-surgical treatment.

DETAILED DESCRIPTION:
The objective of this study is to determine whether enhanced micronutrient intake in the form of fruit, vegetable and berry juice powder (FVB) concentrate, improves clinical outcomes in chronic periodontitis patients prior to non-surgical treatment. In addition, the effects of supplementation prior to and following standard non-surgical management will be assessed, relative to a placebo supplemented group.

The investigators hypothesize that 3-months of nutritional support using this FVB will result in additional reductions in marginal gingival inflammation (bleeding) and additional reductions in probing pocket depth (mean & cumulative), over and above any placebo-related or behavioral effect. In addition, the investigators hypothesize that 3-months of nutritional support prior to a standard non-surgical therapy in conjunction with a continuation of the nutritional support for 3 months will result in further additional reductions in marginal gingival inflammation and probing pocket depth, over and above any placebo-related or behavioral effect following standard non-surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 years old and over
* have a minimum of 20 teeth
* have chronic periodontitis
* be capable of giving informed consent themselves

Exclusion Criteria:

* Patients with aggressive disease
* Patients with physical or mental disability
* Pregnant women or those breastfeeding
* Patients whose medical history may place them at risk of complications from periodontal therapy (e.g. warfarinised Volunteers)
* Patients taking long term anti-microbial or anti-inflammatory drugs
* Patients unable to swallow the study capsules, or take 6 of these capsules a day
* Patients unable to provide informed consent
* Taking dietary supplements (e.g. multivitamins, antioxidants, fish oils) or have taken them within 1-month of the study
* Shows unwillingness, inability or lack of motivation to carry out the study procedures or is not prepared to give written consent or to refrain from using other oral hygiene products (mouthwashes, chewing gum, water piks etc.) or to undergo professional dental cleaning for the duration of the study (other than as part of this protocol)
* Antibiotic or anti-inflammatory therapy currently or in previous two weeks
* Current orthodontic treatment
* Currently participating in another Dental Trial
* Diabetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in clinical parameters | 3 months
  The primary outcomes will be differences in the changes in the below parameters at 3-months post-supplementation between test and placebo groups:
  * % sites with marginal bleeding on probing (BOP) from baseline.
  * Probing pocket depth reductions (mm) from baseline (expressed as reductions in mean and also cumulative pocket depth).
Changes in clinical parameters | 6 months
  The primary outcomes will be differences in the changes in the parameters listed below at 6 months (3 months post supplementation + 3 months post treatment)in test and placebo groups
  % sites with marginal BOP from baseline. Probing pocket depth reductions (mm) from baseline (expressed as reductions in mean and also cumulative pocket depth).

SECONDARY OUTCOMES:
Clinical and biochemical changes | 3 months
  Secondary outcome measures will be clinical and biochemical and include differences in the changes in the below between test and placebo groups:
  * Patient outcomes - oral health quality of life
  * Clinical outcomes - % sites BOP from pocket base from baseline, clinical attachment level (CAL) measures (mm), recession (mm), gingival redness (MGI).
  * Biochemical outcomes in plasma -carbonyls, 8OHdG (from buffy coats), isoprostanes, vitamin C, beta-carotene
Clinical and biochemical changes | 6 months
  Secondary outcome measures will be clinical and biochemical and include differences in the changes in the below between test and placebo groups:
  Patient outcomes - oral health quality of life Clinical outcomes - % sites BOP from pocket base from baseline, CAL measures (mm), recession (mm), gingival redness (MGI).
  Biochemical outcomes in plasma -carbonyls, 8OHdG (from buffy coats), isoprostanes, vitamin C, beta-carotene

CONTACTS AND LOCATIONS:
Overall Officials: Iain L Chapple, BDS, PhD, Principal Investigator — University of Birmingham; Ulrich Schlagenhauf, PhD, Principal Investigator — University of Wuerzburg; Ubele Van der Velden, PhD, Principal Investigator — Academic Centre for Dentistry in Amsterdam
Locations (3):
- University of Wuerzburg, Würzburg, Germany
- Academic Centre for Dentistry, Amsterdam, Netherlands
- Birmingham Dental Hospital & School, Birmingham, West Midlands, United Kingdom